CLINICAL TRIAL: NCT02597439
Title: Placebo-controlled Trial in Subjects at Ultra-high Risk for Psychosis With Omega-3 Fatty Acids in Europe
Acronym: PURPOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rene Kahn (Other)
Responsible Party: Sponsor-Investigator, Rene Kahn, Prof. dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABR54654; 2015-003503-39 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-11-05 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Ultra High Risk for Psychosis
Keywords: Ultra-high risk; UHR; psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acids (Active Comparator): Subjects will be treated daily with 1.2 gram omega-3 polyunsaturated fatty acids (720 mg eicosapentaenoic acid (EPA) and 480 mg Docosahexaenoic acid(DHA)) for six months.
  Interventions: Drug: Omega-3 fatty acids
- Placebo (Placebo Comparator): Subjects will be treated daily with placebo for six months. Placebo capsules will contain a 1:1 combination of coconut oil and medium chain triglycerides because these do not contain polyunsaturated fatty acids and have no impact on omega-3 fatty acid metabolism. Placebo capsules also contain the same amount of vitamin E as the omega-3 capsules and 1% fish oil to mimic flavour and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega-3 fatty acids
  Other Names: Fishoil
  Arms: Omega-3 fatty acids
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether omega-3 fatty acids are effective in the prevention of psychosis in individuals at ultra-high risk for psychosis.

DETAILED DESCRIPTION:
PURPOSE is a randomized double-blind placebo-controlled study. Main objective is to assess the effectivity of omega-3 fatty acid treatment in the prevention of psychosis. The primary outcome measure is the rate of transition to psychosis as determined through CAARMS. Subjects in the age range of 13-20 years with a higher chance of developing psychosis, as determined by the CAARMS, are treated for 6 months with omega-3 fatty acids or placebo. This study in conducted at 14 sites in 9 countries.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject. For individuals younger than 18 years of age the parents / legal representatives need to give consent, and the subject can provide assent (whether the latter is required depends on local laws and regulations).
* UHR diagnosis as made using the Comprehensive Assessment of At-Risk Mental States (CAARMS) (Yung et al., 2005). Subjects have to meet one or more of the following criteria: (a) attenuated psychotic symptoms, (b) brief limited intermittent psychotic symptoms (a history of one or more episodes of frank psychotic symptoms that resolved spontaneously within 1 week in the past year), or (c) either the presence of schizotypal personality disorder or a family history of psychosis in a first-degree relative, all three together with a recent decline in function.

Exclusion Criteria:

* Any clinically significant medical condition that may influence the results of the trial or affect the ability to take part in a trial.
* Laboratory screening values considered clinically relevant by a medical doctor for transaminases, thyroid hormones or coagulation parameters
* Current or past DSM-IV diagnosis of psychosis, as measured with K-SADS-PL
* Current treatment with an antipsychotic or mood-stabilising agent
* Intake of an antipsychotic or mood-stabilising agent in the two weeks prior to study inclusion
* Intake of an antipsychotic agent equivalent to a total haloperidol use of >50 mg in the six months prior to study inclusion
* A first-degree relative (i.e. parents, offspring or siblings) participating in this study
* UHR diagnosis on the basis of attenuated psychotic symptoms that are entirely explained by acute intoxication
* Current aggression or dangerous behaviour (PANSS G14 score 5 or above)
* Current suicidality / self-harm (PANSS G6 score 7)
* Current DSM-IV diagnosis of alcohol or substance dependence as measured with K-SADS-PL
* Any current or previous neurological disorder, including epilepsy
* History of head injury resulting in unconsciousness lasting at least 1 hour
* IQ < 70
* More than 4 weeks of regular omega-3 supplementation (>2 daily capsules standard strength providing >600 mg combined EPA/DHA) within the last 6 months.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Transition rate | 2 years
  To compare transition rates to psychosis during 2 years of follow-up between the omega-3 fatty acids arm and the placebo arm. Starting point is the first administration of medication at the end of visit 2. Endpoint is the moment that a UHR subject makes a transition to psychosis according to the CAARMS criteria.

SECONDARY OUTCOMES:
Discontinuation rate | 2 years
Symptomatology | 2 years
  Symptomatology will be examined with the CAARMS.
Psychosocial functioning | 2 years
  As determined by the Social and Occupational Functioning Assessment Scale (SOFAS)
Cognitive function | 2 years
  Cognitive function is determined by the WAIS
MRI measures | 2 years
  Brain structure and function are measured in three MRI sessions, consisting of structural MRI, resting state functional MRI, Diffusion Tensor Imaging (DTI), and functional MRI during reward processing.
Blood levels of bioactive lipids | 2 years
  Assessment of the omega-3 to omega-6 ratio
Tolerability associated with omega-3 fatty acid treatment | 2 years
  Number of participants with treatment-related adverse events as assessed by the physician.
Blood levels of (epi)genetic markers | 2 years
  Epigenetic markers of interest include but are not restricted to GAD1 and RELN, which are genes coding for the proteins GAD67 and reelin, respectively.
Blood levels of immune parameters | 2 years
  Immune parameters that are assessed include but are not restricted to interferon-γ, interleukin (IL)-1α, IL-1RA, IL-5, IL-10, IL12p40, IL-15, IL-18 and tumour necrosis factor-α.
Positive and negative symptoms | 2 years
  Symptomatology will be examined with the Positive and Negative Syndrome Scale (PANSS).
Level of functioning | 2 years
  Symptomatology will be examined with the Global Assessment of Functioning scale (GAF).
Clinical Impression | 2 years
  Symptomatology will be examined with the Clinical Global Impression Scale (CGI).
Level of depression | 2 years
  Symptomatology will be examined with the Beck's Depression Inventory (BDI).
Role functioning | 2 years
  Determined by the Global Functioning Role (GF:R) scale
Social functioning | 2 years
  Determined by the Global Functioning Social (GF:S) scale.

CONTACTS AND LOCATIONS:
Overall Officials: René Kahn, Prof. Dr., Study Chair — UMC Utrecht
Locations (14):
- BioPsyC Biopsychosocial Corporation, Vienna, Austria
- Department of Child and Adolescent Psychiatry, University of Tübingen, Tübingen, Germany
- Israel (2):
  - Schneider Children's Medical Center, Petah Tikva
  - Tel Hashomer The Sheba Medical Center, Ramat Gan
- Italy (2):
  - Fondazione Santa Lucia, Rome
  - Sapienza University of Rome, Rome
- Brain Center Rudolf Magnus, Department of Psychiatry, University Medical Center Utrecht, Utrecht, Netherlands
- Institute of Clinical Medicine, University of Bergen, Bergen, Norway
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Infantil Passeig Sant Joan de Deu, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Idival, University of Cantabria, Cibersam Unidad de investigacion en psiquiatria, Santander
- ZKJP University Zürich, Zurich, Switzerland
- Psychiatry, Centre for Clinical Brain Sciences, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Winter-van Rossum I, Slot MIE, van Hell HH, Bossong MG, Berger G, Aschauer H, Maat A, Walitza S, Lavan O, Baeza I, Dolz M, Monducci E, Fiori Nastro P, Kroken RA, Lawrie SM, Diaz-Caneja CM, Renner T, Schlogelhofer M, Scharinger C, Spalletta G, Banaj N, Otero S, Schipper M, Kwakkel DB; PURPOSE Study Group; Kahn RS. Effectiveness of Omega-3 Fatty Acids Versus Placebo in Subjects at Ultra-High Risk for Psychosis: The PURPOSE Randomized Clinical Trial. Schizophr Bull. 2025 Jul 7;51(4):1082-1091. doi: 10.1093/schbul/sbae186. PMID 39450759